CLINICAL TRIAL: NCT03202030
Title: Immediate Dentoalveolar Restoration Compared to Demineralized Bovine Bone in Immediate Implants Placed in Fresh Sockets With Buccal Bone Resorption: 18-months Randomized Controlled Trial
Brief Title: Immediate Dentoalveolar Restoration Compared to Bio-oss
Acronym: IDRBio-oss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: University of the Republic, Uruguay (Other)
Responsible Party: Principal Investigator, Alex Nogueira Haas, Professor, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Udelar
Record Dates: First submitted 2017-06-26; First posted 2017-06-28 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Fresh Sockets With Buccal Resorption
Keywords: immediate dentoalveolar restoration; bio-oss; immediate dental implant; bovine bone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDR (Experimental): Immediate dentoalveolar restoration conducted with bone removed from the tuber
  Interventions: Procedure: Immediate dentoalveolar restoration
- Bio-oss (Active Comparator): Bovine demineralized bone (Bio-oss Collagen) applied on the buccal resorption of the immediate implant
  Interventions: Procedure: Demineralized bovine bone

INTERVENTIONS:
Procedure: Immediate dentoalveolar restoration — Block of bone removed from the tuber and placed in the buccal resorption of the socket together with an immediate implant
  Other Names: IDR
  Arms: IDR
Procedure: Demineralized bovine bone — Block of demineralised bovine bone placed in the buccal resorption of the socket together with an immediate implant
  Arms: Bio-oss

SUMMARY:
This randomised controlled trial compares the immediate dentoalveolar restoration and bovine demineralised bone in immediate implants placed in fresh sockets with buccal resorption. A total of 34 patients will be included and followed clinically and radiographically for 18 months. Patient centred outcomes will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Tooth extraction indicated for teeth in anterior area between second premolars

Exclusion Criteria:

* Diabetes and other systemic conditions that may affect osseointegration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Buccal-palatal thickness | 18 months

SECONDARY OUTCOMES:
Oral-health related quality of life | 18 months
  The OHIP-14 will be applied and satisfaction will also be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de La Republica del Uruguay, Montevideo, Uruguay

IPD SHARING:
Plan to Share IPD: No